CLINICAL TRIAL: NCT03934294
Title: Acupuncture Effect on Digestion in Critically Ill Post-Operative Oral and Hypo-pharyngeal Cancer Patients: A Protocol for Double Blind Randomized Control Trial
Brief Title: Acupuncture Effect on Digestion in Critically Ill Post-Operative Oral and Hypo-pharyngeal Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMUH108-REC2-037(AR-1)
Record Dates: First submitted 2019-04-28; First posted 2019-05-01 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Oral Cancer; Hypopharyngeal Cancer
Keywords: Critically ill; Intensive care; Oral cancer; Hypo-pharyngeal cancer; Acupuncture; Digestion; ICU
MeSH Terms: conditions — Mouth Neoplasms; Hypopharyngeal Neoplasms; Critical Illness | interventions — Metoclopramide

STUDY DESIGN:
Intervention Model Description: two groups, randomized, pre-post intervention study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients will be randomized to one of two groups: Acu/ Con in a 1:1 ratio. The random number and patient name will be written down on an non transparent envelope by a study nurse. The study nurse will provide an envelope containing a sheet depicting the acupoint name, location and picture (Acu / Con) to the acupuncture doctor. Acupuncture doctor (blind) will preform acupuncture on the points. 30 minutes after needle insertion, acupuncture doctor will withdraw the needles. Acupuncturists, ICU nurses, ICU doctors, researchers and statisticians will all be blind to group allocation and to the meaning of the random numbers until all acupuncture treatments have been completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group: specific acupuncture group(Acu) (Experimental): In addition to routine ICU treatments, patients in the specific acupuncture group will also receive daily bilateral traditional Chinese medicine style acupuncture on the following acupuncture points: ST36 (Zu San Li), ST37 (Shangjuxu), ST39 (Xiajuxu), PC6 (Nei Guan) and LI4 (He Gu). The acupoints indications in this group are specific to treat indigestion related conditions. The treatment will take place once a day, over three days, for a total of three treatments. A total of 10 Needles will be used in each session Acupuncture treatment will be performed with sterile needles manufactured by "Yu Kuang" acupuncture needles 40mm with 30G.
  Acupuncture doctor will disinfect the acupoints with alcohol and will perform acupuncture on the marked points with needle Needle retention time will be 30 minutes. The needles will be withdrawn by acupuncture doctor.
  Interventions: Other: Specific acupuncture group; Drug: Metoclopramide 10mg
- Control group: non-specific acupuncture group (Con-Acu) (Placebo Comparator): Patients' in the non-specific acupuncture group (Con-Acu) will receive routine ICU treatment as well as a total of 3 daily non digestion related Traditional Chinese medicine style acupuncture treatments at the following acupoints: LI 15 (Jianyu), SJ 14 (JianLiao) LU3 (Tianfu), GB35 (Yangjiao), BL 59 (Fuyang). The selected control points are not indicated for the treatment of digestion related pathologies, and are not reported to improve digestive function.
  Acupuncture doctor 1 will disinfect the marked acupoints with alcohol and will perform acupuncture on the marked points. Needle retention time will be 30 minutes. The needles will be withdrawn by acupuncture doctor
  Interventions: Drug: Metoclopramide 10mg; Other: Non-specific acupuncture group

INTERVENTIONS:
Other: Specific acupuncture group — In addition to routine ICU treatments, patients in the specific acupuncture group will also receive daily bilateral traditional Chinese medicine style acupuncture on the following acupuncture points: ST36 (Zu San Li), ST37 (Shangjuxu), ST39 (Xiajuxu), PC6 (Nei Guan) and LI4 (He Gu). The acupoints indications in this group are specific to treat indigestion related conditions. The treatment will take place once a day, over three days, for a total of three treatments. A total of 10 Needles will be used in each session Acupuncture treatment will be performed with sterile needles manufactured by "Yu Kuang" acupuncture needles 40mm with 30G.
  Other Names: Specific acupuncture to treat indigestion
  Arms: Treatment group: specific acupuncture group(Acu)
Drug: Metoclopramide 10mg — Patients in all groups will receive Metoclopramide 10mg/ per 8 hours in the case of poor digestion, alongside the individualized drug treatment prescribed by the ICU medical doctor as per individual patient needs.
  Other Names: Metoclopramide 10mg/ per 8 hours in the case of poor digestion
Other: Non-specific acupuncture group — Patients' in the non-specific acupuncture group (Con-Acu) will receive routine ICU treatment as well as a total of 3 daily non digestion related Traditional Chinese medicine style acupuncture treatments at the following acupoints: LI 15 (Jianyu), SJ 14 (JianLiao) LU3 (Tianfu), GB35 (Yangjiao), BL 59 (Fuyang). The selected control points are not indicated for the treatment of digestion related conditions, and are not reported to improve digestive function.
  Other Names: Non specific acupuncture to treat indigestion
  Arms: Control group: non-specific acupuncture group (Con-Acu)

SUMMARY:
Background: Head and neck cancer patients are in high risk to suffer from malnourishment, a risk that increase in postoperative condition and with the use of enteral nutrition (EN). Until now patients who are suffering from indigestion in the ICU received treatment in the form of prokinetic drugs, drags that can lead to serious side effects and only can partially improve digestion. Acupuncture was used successfully in several clinical trials to improve postoperative indigestion in cancer patients without any reported adverse events. This study aims is to design a double blind settings in order to investigate acupuncture effect in combination of prokinetic drugs in the prevention of indigestion in postoperative oral and hypo-pharyngeal cancer patients in the Intensive Care Unit (ICU).

Methods: Single center, double blind randomize control trial will compare between two equal groups. A total of 28 patients that will meet the inclusion criteria: Age 30-80, Post plastic surgery for oral cancer or hypo-pharyngeal cancer, Apache score below 20 needed EN. Patients will be randomly divided into specific acupuncture (ACU) or non-specific acupuncture (CON) for 3 treatments in 3 days by a blind acupuncturist along with prokinetic drugs. The main outcome measurement will be the amount of days a patient need to reach Total Energy Expenditure (TEE).

Expected outcome: The results will shed light on the effectiveness and safety of acupuncture in a double blind design for posts-surgery ICU cancer patients. In addition, the study presents a revolutionary double blind design that if will prove as successful might influence the way double blind acupuncture studies are performed today.

DETAILED DESCRIPTION:
Background: Head and neck cancer patients are in high risk to suffer from malnourishment, a risk that increase in postoperative condition and with the use of enteral nutrition (EN). Until now patients who are suffering from indigestion in the ICU received treatment in the form of prokinetic drugs, drags that can lead to serious side effects and only can partially improve digestion. Acupuncture was used successfully in several clinical trials to improve postoperative indigestion in cancer patients without any reported adverse events. This study aims is to design a double blind settings in order to investigate acupuncture effect in combination of prokinetic drugs in the prevention of indigestion in postoperative oral and hypo-pharyngeal cancer patients in the Intensive Care Unit (ICU).

Methods: Single center, double blind randomize control trial will compare between two equal groups. A total of 28 patients that will meet the inclusion criteria: Age 30-80, Post plastic surgery for oral cancer or hypo-pharyngeal cancer, Apache score below 20 needed EN. Patients will be randomly divided into specific acupuncture (ACU) or non-specific acupuncture (CON) for 3 treatments in 3 days by a blind acupuncturist along with prokinetic drugs. The main outcome measurement will be the amount of days a patient need to reach his Total Energy Expenditure (TEE).

Expected outcome: The results will shed light on the effectiveness and safety of acupuncture in a double blind design for posts-surgery ICU cancer patients. In addition, the study presents a revolutionary double blind design that if will prove as successful might influence the way double blind acupuncture studies are performed today.

Other information: The study will be conducted in the surgical ICU department, of china medical university hospital, Taichung 404, Taiwan. The study in conducted on stable ICU patients and is anticipated to have a minimum risk for adverse events. Patients enrollment and data collection will start immediately after china medical hospital research ethics committee approval. The study expected completion time: June 2021

ELIGIBILITY:
Inclusion Criteria:

* Age 30-80
* Apache score below 20
* Patients needed EN
* Post plastic surgery, including oral cancer or hypo-pharyngeal cancer

Exclusion Criteria:

* Coagulopathy,
* prolong prothrombin time (PPT) activated partial thromboplastin time (aPTT) more then 4 times
* Thrombocytopenia - low platelet count
* Clinically unstable: receiving two inotropic agents or Fraction of inspired Oxygen (FiO2) >70%
* Estimated ICU stay - less than 3 days

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2021-03-19 (Actual); Study Completion 2021-03-19 (Actual)

PRIMARY OUTCOMES:
Time to reach Total Energy Expenditure | Up to 1 month
  Number of days in takes for each patient to achieve the Total Energy Expenditure

SECONDARY OUTCOMES:
Amount of prokinetic drugs prescribed | Up to 1 month
  Secondary outcomes measures are the amount of prokinetic drugs prescribed by the ICU doctor in total dosage
The need of naso-jejunal feeding tube | Up to 1 month
  After 5 days of conservative treatment for the poor digestion (naso-gastric tube drainage of more than 500ml per day or severe diarrhea of more than 1000 ml per day)
The need of parental nutrition | up to 1 month
  In patients who cannot digest with daily naso-gastric tube drainage of more than 500ml per day or severe diarrhea of more than 1000 ml per day
Incidents of vomits | Up to 1 month
  Incidents of vomits in total number of times and volume in micro liters
Albumin blood levels | Up to 1 month
  Patient's Albumin blood levels will help to assets patient's nutrition status
Total ICU stay | Up to 23 month
  Total ICU stay in days
Total hospital stay | Up to 23 month
  Total hospital stay in days
Total mechanical ventilation in days | Up to 23 month
  A day of mechanical ventilation is at least 6 hours of mechanical ventilation in one day
Total mortality | Up to 23 month
  In case of mortality ,total mortality will be compered between the two groups
Incidents of diarrhea | Up to 1 month
  Incidents of diarrhea in number of times and volume in micro liters
Incidents of constipation | Up to 1 month
  No stool passage in 3 days will be considered as constipation
Incidents of nausea | Up to 1 month
  Incidents of nausea in number of times , measured by patient complains
Incidents of gastrointestinal bleeding | Up to 1 month
  Positive occult blood test of the naso-gastric tube drainage and in the stool
Incidents of fever episodes | Up to 1 month
  Body temperature more than 38 degrees Celsius

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Yu Kao, M.D., Principal Investigator — China Medical University Hospital
Locations (1):
- surgical and burn intensive care departments and the plastic surgical department of China Medical University Hospital in Taichung city, Taiwan., Taichung, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No